CLINICAL TRIAL: NCT07171905
Title: Exploring the Role of Carbonic Anhydrase IX as Diagnostic and Theranostic Target in Von-hippel Lindau Disease
Brief Title: CAT-VHL Exploring the Role of Carbonic Anhydrase IX as Diagnostic and Theranostic Target in Von-Hippel Lindau Disease
Acronym: CAT-VHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Larcher Alessandro, Medical Doctor, IRCCS Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNRR-POC-2023-12377493
Record Dates: First submitted 2025-03-25; First posted 2025-09-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: VHL - Von Hippel-Lindau Syndrome
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Intervention Model Description: phase 2, non-comparative and non-randomized, single arm, open-label, multicenter, national, no-profit clinical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- investigating the role of CAIX as target in VHL disease and in VHL-/- tumors (Experimental)
  Interventions: Drug: investigating the role of CAIX as target in VHL disease and in VHL-/- tumors.

INTERVENTIONS:
Drug: investigating the role of CAIX as target in VHL disease and in VHL-/- tumors. — Participants VHL disease and in VHL-/- tumors, will receive a single dose of the diagnostic radiopharmaceutical [89Zr]Zr-DFO-Girentuximab and subsequently undergo imaging with a hybrid PET/CT scanner.

SUMMARY:
The study is a phase 2, non-comparative and non-randomized, single arm, national clinical trial testing the hypothesis that CAIX-PET has diagnostic and theranostic potential in VHL disease and in VHL-/- tumors. Participants will receive a single dose of the diagnostic radiopharmaceutical [89Zr]Zr-DFO-Girentuximab and subsequently will be subjected to imaging with an hybrid PET/CT scanner. Sensitivity and diagnostic accuracy of experimental imaging will be assessed against standard of truth derived from standard of care procedures such as MRI or pathology following surgery. A theranostic approach will be simulated by replacing the physical decay of the diagnostic isotope [89Zr]Zr with the physical decay of therapeutic isotopes and evaluating tissue dosimetry.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily given informed consent
* Age ≥18 years old
* Performance Status ECOG/WHO score 0-2
* For females of reproductive potential, negative pregnancy test and use of highly effective contraception for 30 days following IMP administration
* For males of reproductive potential, use of highly effective contraception for 30 days following IMP administration.

And, for the primary cohort:

* Diagnosis of VHL disease requiring surveillance following confirmation of pathogenic variant at genetic test

Alternatively, for the secondary cohort:

- Clinical and/or pathological diagnosis of hemangioblastoma, pheochromocytoma, pancreatic neuroendocrine tumor or clear cell renal cell carcinoma requiring surgery.

Exclusion Criteria:

* Performance Status ECOG/WHO score >2
* Women who are pregnant or breastfeeding or are planning pregnancy during the study
* Men who are planning fatherhood during the study
* Exposure to any murine or chimeric antibodies within 5 years prior to the planned IMP administration
* Exposure to any experimental diagnostic or therapeutic drug within 30 days from the planned IMP administration
* Surgery, biopsy, ablative procedure, radiotherapy or any other local treatment for any primary tumor within 4 weeks prior to the planned IMP administration
* Exposure to any systemic agent within 4 weeks prior to the planned IMP administration or in case of continuing adverse effects with grade >1 from such therapy
* Current exposure to systemic agents or scheduled therapy in the next 6 months following the planned IMP administration
* Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic) that may interfere with the objectives of the study or within the safety of compliance of the subjects as judged by the Investigator
* Known hypersensitivity to [89Zr]Zr-DFO-Girentuximab or DFO (Desferrioxamine)
* Severe chronic kidney disease with glomerular filtration rate ≤ 30 mL/min/1.73m2
* Other vulnerable categories than rare disease (e.g, being in detention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
to assess the efficacy of CAIX-PET | IMP administration at day 0; CAIX-PET from day 3 to 7; MRI according to standard of care and imaging assessment from day 1 to 60.
  to assess the Sensitivity of CAIX-PET for the diagnosis of tumors in VHL disease

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italia, Italy